CLINICAL TRIAL: NCT01776099
Title: Diabetes Nutrition Algorithms - Sugars: Galactose- and Fiber-induced Metabolic Improvement in the Dietetic Treatment of Type 2 Diabetes
Acronym: DiNA-S DiNA-F
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Firma Rettenmeier & Söhne (Company) (Unknown); German Center for Diabetes Research (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Director of the Department for Clinical Nutrition, German Institute of Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DiNA-S DiNA-F
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; nutrition; fibers
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- pure galactose (Active Comparator): 5 grams of galactose, three times a day with the main meals, duration: 4 weeks
  Interventions: Dietary Supplement: Dietary supplement (4 arms, 2 active, 2 placebo)
- pure palatinose (Placebo Comparator): 5 grams of palatinose, three times a day with the main meals, duration: 4 weeks
  Interventions: Dietary Supplement: Dietary supplement (4 arms, 2 active, 2 placebo)
- soluble non-fermentable fibers (Placebo Comparator): 5 grams of soluble non-fermentable fibers, three times a day with the main meals, duration: 4 weeks
  Interventions: Dietary Supplement: Dietary supplement (4 arms, 2 active, 2 placebo)
- non-soluble non-fermentable fibers (Active Comparator): 5 grams of non-soluble non-fermentable fibers, three times a day with each main meal, duration: 4 weeks
  Interventions: Dietary Supplement: Dietary supplement (4 arms, 2 active, 2 placebo)

INTERVENTIONS:
Dietary Supplement: Dietary supplement (4 arms, 2 active, 2 placebo)

SUMMARY:
In animal models and retrospective studies, certain food components such as sugars and fiber have been detected as potential agents to influence development and progress of type 2 diabetes.

The DiNA study prospectively investigates, if non-soluble non-fermentable fibers (vs. soluble ones) and galactose (vs. palatinose) are capable to improvement metabolic parameters in patients with long-term type 2 diabetes and intensive insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes, insulin-dependent
* high insulin resistance

Exclusion Criteria:

* accompanying disease, medication or metabolic disorder, which interact with glucose metabolism or eating behavior (e.g. renal insufficiency, major cardial insuffiency, untreated hypothyreosis, corticoid treatment, depression and other psychiatric disorders...)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
metabolic improvement of type 2 diabetes | 4 weeks
  metabolic improvement of type 2 diabetes, as to be shown via hyperinsulinemic-euglycaemic clamp, mixed-meal test and daily demand of insulin units

CONTACTS AND LOCATIONS:
Overall Officials: Andreas F.H. Pfeiffer, Prof. Dr. med., Principal Investigator — German Institute for Human Nutrition
Locations (1):
- Charité-Klinikum Benjamin Franklin, Berlin, Germany